CLINICAL TRIAL: NCT05480046
Title: Risperidone ISM® Effectiveness in Schizophrenia Patients Hospitalised Due to A Relapse: a Prospective Non-interventional Evaluation (RESHAPE Study)
Brief Title: Non-interventional Study of Risperidone ISM® in Schizophrenia Patients Hospitalised Due to a Relapse
Acronym: RESHAPE
Status: Completed | Type: Observational
Sponsor: Rovi Pharmaceuticals Laboratories (Industry)
Responsible Party: Sponsor
Other Study IDs: ROV-RISP-2021-01
Record Dates: First submitted 2022-07-20; First posted 2022-07-29 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Schizophrenia
Keywords: Risperidone; Schizophrenia; Long-acting injectable
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Drug: Risperidone ISM — Risperidone ISM is administered every 4 weeks
  Other Names: OKEDI®

SUMMARY:
This is a prospective, non-interventional, multicentre study designed to collect information about the effectiveness, safety and tolerability of Risperidone ISM in patients diagnosed with schizophrenia who are suffering an acute exacerbation, according to routine clinical practice.

DETAILED DESCRIPTION:
This is a non-interventional, multicentre, prospective study conducted in psychiatric inpatient units, and designed to collect information about the effectiveness, safety and tolerability of Risperidone ISM in patients diagnosed with schizophrenia and who are suffering an acute exacerbation, according to routine clinical practice.

The study comprises five visits in total:

Baseline Visit: This visit must be conducted within 48 hours after the first injection of Risperidone ISM. During this visit, the patient must meet all inclusion and exclusion criteria and sign the Informed Consent Form.

Follow-up Visit I: Scheduled approximately 8 ± 2 days after the first injection.

Follow-up Visit II: Scheduled approximately 28 ± 2 days after the first injection.

Discharge Visit: Conducted on the day of discharge, which may vary depending on the individual patient.

Final Visit: Occurs approximately 28 days after the second injection of Risperidone ISM and may be conducted in person or via telephone.

The study will be conducted in five visits: the Baseline Visit is the day on which the patient fulfils the inclusion and exclusion criteria, including signature of the Informed Consent; two follow-up visits will be scheduled after the first injection of Risperidone ISM; in addition, there will be another visit on the day of discharge; and the Final Visit will occur approximately 28 days after the 2nd injection of Risperidone ISM.

The primary objective of the study is to assess, under usual clinical practice, the effectiveness of Risperidone ISM in patients hospitalised due to a schizophrenia relapse.

The secondary objectives include:

Analysis of patterns of use of Risperidone ISM in hospital settings across several European countries.

Characterisation of patient profiles treated with Risperidone ISM in routine clinical practice.

Assessment of social functioning in schizophrenia patients treated with Risperidone ISM.

Evaluation of duration of hospitalisation across participating countries. Measurement of patient-reported treatment satisfaction. Evaluation of safety and tolerability of Risperidone ISM in routine clinical practice.

To assess these objectives, the following scales will be used:

PANSS-6: Baseline visit, Follow-up Visit I, Follow-up Visit II, and Final Visit.

CGI-S: Baseline visit, Follow-up Visit I, Follow-up Visit II, and Final Visit. PSP: Baseline visit, Follow-up Visit II, and Final Visit. MSQ: Baseline visit, Follow-up Visit II, and Final Visit.

Approximately 1,200 adults' patients were calculated to be enrolled in the sites from the participating countries.

The initial sample size estimation relied on an extremely small effect size that would be very unlikely given the results on a previous clinical trial with Risperidone ISM. After the examination of preliminary trial data and considering that the recruitment period was going to be longer than expected (mostly related to administrative issues for activating sites), the Sponsor has decided to re-evaluate the sample size required for the study. For this new estimation, the objective was to calculate the sample size that would allow to perform the analyses of the primary effectiveness variables not only in the total study population, but also in the subgroups who were pre-specified in the study protocol. Accordingly, the estimation was adjusted for each of the subgroups estimated share of the total study sample, and then accounted for the expected loss of patients, that was adjusted upwards to 35%. After that, the new sample size was set at approximately 272 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged 18 years or older at the time of hospitalisation.
2. Patient with diagnosis of schizophrenia, as per clinical judgment.
3. Patient admitted to a psychiatric inpatient unit due to an acute exacerbation.
4. Patient has started treatment with Risperidone ISM within the previous 48 hours, according to the current Summary of Product Characteristics (SmPC).
5. Patient or their legal representative provides written informed consent to participate in the study.

Exclusion Criteria:

1. Patient with a diagnosis of schizoaffective disorder, bipolar disorder mental retardation, or other cognitive and neurodevelopmental disorders.
2. Patient with substance-induced psychosis or psychosis during intoxication (patients with comorbid substance abuse/dependence are allowed).
3. Patient unable to answer the study questionnaires.
4. Patient who is currently participating in another clinical study.
5. Patient pregnant or breast-feeding.
6. Patient with a serious and unstable medical condition, forensic patients, or patients with any contraindication mentioned in the SmPC of Risperidone ISM.
7. Patients currently on antipsychotic treatment with clozapine or any long-acting injectable antipsychotic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 diagnosed with schizophrenia who are admitted to a psychiatric unit due to a relapse and initiate treatment with Risperidone ISM (OKEDI®), according to the therapeutic indication of the marketing authorization ("Treatment of schizophrenia in adults for whom tolerability and effectiveness has been established with oral risperidone") under routine clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 275 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2025-03-13 (Actual); Study Completion 2025-03-13 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impression-Severity of Illness scale (CGI-S): change from baseline to Day 56. | Baseline and Day 56 (or the last post-baseline assessment)
  The Clinician Global Impression - Severity (CGI-S) score is a 7-point clinician-rated scale for assessing the global severity of the illness. A rating of 1 is equivalent to "Normal, not at all ill" and a rating of 7 is equivalent to "Among the most extremely ill participants". Negative change from baseline scores indicate improvement in the severity of illness whereas higher scores mean a worse outcome.
Positive and Negative Syndrome Scale (PANSS-6): change from baseline to Day 56. | Baseline and Day 56 (or the last post-baseline assessment)
  The six-item version of the Positive and Negative Syndrome Scale (PANSS-6) is a 6-item scale derived from the full 30-item PANSS which evaluate: Delusions, Conceptual disorganization, Hallucinations, Blunted Affect, Social withdrawal and Lack of spontaneity and flow of conversation Safety and tolerability.

SECONDARY OUTCOMES:
Personal and Social Performance (PSP) scale | Baseline and Day 56 (or the last post-baseline assessment)
  The PSP is a 100-point single-item rating scale that is based on 4 areas: personal and social relationships; self-care; work and socially useful activities, and disturbing and aggressive behaviors. Each of the 4 domains is rated in 6 degrees of severity (absent, mild, manifest, marked, severe, very severe). Higher PSP scores indicate a better social functioning.
Medication Satisfaction Questionnaire (MSQ) | Day 56 (or the last post-baseline assessment)
  The Medication Satisfaction Questionnaire (MSQ) is a single-item, global, patient-completed instrument designed to assess treatment satisfaction among patients with schizophrenia. It consists of 1 question: "Overall, how satisfied are you with your current antipsychotic medication(s)?" with responses assessed on a 7-point scale rated as follows: 1 = extremely dissatisfied, 2 = very dissatisfied, 3 = somewhat dissatisfied, 4 = neither satisfied nor dissatisfied, 5 = somewhat satisfied, 6 = very satisfied, 7 = extremely satisfied.
Duration of hospitalisation | Baseline and Day 56 (or the last post-baseline assessment)
  The duration of hospitalisation is the time from admission in the hospital to discharge.
Adverse drug reactions (ADR) | Up to Day 56 (or the last post-baseline assessment)
  An adverse drug reaction (ADR), is a response to a study treatment that is noxious and unintended and that occurs at doses normally used in man for prophylaxis, diagnosis or therapy of disease, or for the restoration, correction, or modification of physiological functions. Response in this context means that a causal relationship between a medicinal product and an adverse event is at least a reasonable possibility.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph U Correll, Study Chair — Charite University, Berlin, Germany
Locations (77):
- Germany (21):
  - Investigational site number DE-06, Aachen
  - Investigational site number DE-14, Ansbach
  - Investigational site number DE-23, Bayreuth
  - Investigational site number DE-10, Berlin
  - Investigational site number DE-12, Berlin
  - Investigational site number DE-15, Berlin
  - Investigational site number DE-07, Bonn
  - Investigational site number DE-16, Bonn
  - Investigational site number DE-02, Chemnitz
  - Investigational site number DE-03, Dortmund
  - Investigational site number DE-25, Eberswalde
  - Investigational Site number DE-01, Essen
  - Investigational site number DE-08, Greifswald
  - Investigational site number DE-22, Hamburg
  - Investigational site number DE-20, Hemer
  - Investigational site number DE-19, Leipzig
  - Investigational site number DE-05, Mannheim
  - Investigational site number DE-04, Munich
  - Investigational site number DE-09, München
  - Investigational site number DE-24, Neustadt
  - Investigational site number DE-13, Werneck
- Italy (15):
  - Investigational site number IT-32, Ancona
  - Investigational site number IT-19, Bolzano
  - Investigational site number IT-24, Brescia
  - Investigational site number IT-65, Brindisi
  - Investigational site number IT-20, Crema
  - Investigational site number IT-41, Foggia
  - Investigational site number IT-03, Legnano
  - Investigational site number IT-47, Manfredonia
  - Investigational site number IT-06, Milan
  - Investigational site number IT-42, Milan
  - Investigational site number IT-18, Montichiari
  - Investigational site number IT-113, Palermo
  - Investigational site number IT-44, Putignano
  - Investigational site number IT-97, Sant'Agata di Militello
  - Investigational site number IT-90, Vimercate
- Portugal (10):
  - Investigational site number PT-25, Beja
  - Investigational site number PT-24, Braga
  - Investigational site number PT-01, Coimbra
  - Investigational site number PT-33, Funchal
  - Investigational site number PT-36, Funchal
  - Investigational site number PT-20, Guarda
  - Investigational site number PT-32, Portimão
  - Investigational site number PT-13, Porto
  - Investigational site number PT-11, Santo Tirso
  - Investigational site number PT-27, Tomar
- Spain (30):
  - Investigational site number ES-03, Barcelona
  - Investigational site number ES-45, Barcelona
  - Investigational site number ES-81, Barcelona
  - Investigational site number ES-16, Burgos
  - Investigational site number ES-23, Córdoba
  - Investigational site number ES-11, Granada
  - Investigational site number ES-59, Huesca
  - Investigational site number ES-21, Jaén
  - Investigational site number ES-70, Jerez de la Frontera
  - Investigational site number ES-72, L'Hospitalet de Llobregat
  - Investigational site number ES-60, Las Palmas de Gran Canaria
  - Investigational site number ES-49, Lleida
  - Investigational site number ES-51, Lugo
  - Investigational site number ES-19, Madrid
  - Investigational site number ES-24, Madrid
  - Investigational site number ES-66, Madrid
  - Investigational site number ES-63, Majadahonda
  - Investigational site number ES-04, Manacor
  - Investigational site number ES-73, Manresa
  - Investigational site number ES-65, Mataró
  - Investigational site number ES-14, Móstoles
  - Investigational site number ES-18, Murcia
  - Investigational site number ES-52, Ourense
  - Investigational site number ES-62, Ponferrada
  - Investigational site number ES-69, Santander
  - Investigational site number ES-02, Talavera de la Reina
  - Investigational site number ES-42, Torrejón
  - Investigational site number ES-76, Úbeda
  - Investigational site number ES-31, Vigo
  - Investigational site number ES-40, Vitoria-Gasteiz
- Investigational site number GB-08, London, United Kingdom